CLINICAL TRIAL: NCT00789438
Title: The Effects of Sedation and Analgesia on the Surgical Pleth Index (SPI)
Brief Title: Evaluation of the Surgical Pleth Index During Spinal and General Anesthesia
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Berthold Bein, Institut für Anästhesiologie und Operative Intensivmedizin, Campus Kiel
Other Study IDs: SSI-154-02
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Results first posted 2010-02-19 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2009-10

CONDITIONS: Stress; Pain
Keywords: Analgesia; Sedation; Spinal; Stress; Surgical; Surgical Stress; Pain
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- General Anesthesia: Patients undergoing short-term surgery (30-90 min) under general anesthesia
- Spinal: Patients undergoing short-term surgery (30-90 min) under spinal anesthesia
- Spinal + Sedation: Patients undergoing short-term surgery (30-90 min) under spinal anesthesia with sedation

SUMMARY:
The Surgical Pleth index (SPI) has been introduced as a non invasive tool to "measure" stress and pain during surgery. Preliminary studies were performed in patients under general anaesthesia with propofol and remifentanil. These trials showed a good correlation between SPI and aching procedures and a negative correlation between SPI and the remifentanil dosage. Hence, it was concluded that SPI may be a bedside tool to measure 'pain' during surgery. So far, no study investigated SPI during regional anaesthesia.

DETAILED DESCRIPTION:
1. Spinal anaesthesia secures full pain relieve and muscle relaxation usually in the lower part of the body. Thus, SPI - a measure that reflects pain during surgery - may not exceed significantly compared to baseline. It may slightly increase only during administration of the block.
2. Increasing SPI values due to surgery under subarachnoid block may reflect intraoperative patient's stress mediated by activation of the autonomic nervous system, specifically sympathetic activation.
3. In consistence with previously published data no changes of SPI should occur due to standardized sedation with propofol.

ELIGIBILITY:
Inclusion Criteria:

* surgical procedures feasible under general or spinal anesthesia
* duration between 30 and 90 min
* ASA status I,II or III

Exclusion Criteria:

* contraindications against one of the anesthesia methods
* age under 18
* emergencies
* chronical pain history
* lack of sinus rhythm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for short-term (30-90 min) surgery.
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2008-10; Primary Completion 2010-01 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Bein, PD Dr med, Study Director — Institut für Anästhesiologie und operative Intensivmedizin, Universitätsklinikum Schleswig-Holstein, Campus Kiel
Locations (1):
- Institut für Anästhesiologie und Operative Intensivmedizin, Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | General Anesthesia | Spinal | Spinal + Sedation
Started | 21 | 20 | 28
Completed | 21 | 20 | 28
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | General Anesthesia | Spinal | Spinal + Sedation | Total
Number analyzed (Participants) | 21 | 20 | 28 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 15 | 21 | 52
  >=65 years | 5 | 5 | 7 | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 59 (16) | 61 (18) | 62 (17) | 60 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 23 | 56
  Male | 5 | 3 | 5 | 13
Region of Enrollment [Number; unit: participants]
  Germany | 21 | 20 | 28 | 69

OUTCOME MEASURES:

1. Primary Outcome: Difference Between All Groups for the Surgical Pleth Index(SPI) at Defined Timepoints
Description: Surgical Pleth Index (SPI), derived from finger photoplethysmographic signal has a range from 0 showing the lowest stress level to 100 showing the maximum stress level. SPI was compared between the groups during six defined time points: baseline (BL)- day before surgery; induction (IND)-before induction of general anesthesia or before spinal punction respectively; intubation (INT) or spinal punction (SPA); skin incision (INC), surgical suture (SU) and 10 minutes after admission to the recovery room (PACU). Difference between the groups is calculated using ANOVA.
Time Frame: Time points for outcome measures: Baseline, before Induction of anesthesia, during Intubation or Spinal Punction, during Skin Incision, during Surgical Suture, during Post Anesthesia Care Unit stay
Measure: Median (Standard Error); unit: SPI and delta SPI (to baseline)
Arm/Group | General Anesthesia | Spinal | Spinal + Sedation
Number analyzed (Participants) | 21 | 20 | 28
SPI and delta SPI (to baseline)
  Median SPI at skin incision | 46 (4) | 67 (3) | 40 (47)

ADVERSE EVENTS:
Arm/Group | General Anesthesia | Spinal | Spinal + Sedation
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/28
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes